CLINICAL TRIAL: NCT03339297
Title: A Phase 2, Prospective, Randomized, Open-Label Study on the Efficacy of Defibrotide Added to Standard of Care Immunoprophylaxis for the Prevention of Acute Graft-versus-Host-Disease in Adult and Pediatric Patients After Allogeneic Hematopoietic Stem Cell Transplant
Brief Title: An Open-Label Study of Defibrotide for the Prevention of Acute Graft-versus-Host-Disease (AGvHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JZP963-201
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Results first posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-07

CONDITIONS: Graft-versus-host Disease; Acute-graft-versus-host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — defibrotide; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Defibrotide Prophylaxis (Experimental): Standard of Care Immunoprophylaxis + Defibrotide
  Interventions: Drug: Defibrotide; Drug: Standard of Care
- Standard of Care (Active Comparator): Standard of Care Immunoprophylaxis Alone
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Defibrotide — 6.25 mg/kg via 2-hour IV infusion every 6 hours
  Arms: Defibrotide Prophylaxis
Drug: Standard of Care — Administered according to local institutional guidelines, physician preference, and patient need.

SUMMARY:
This is a study comparing the defibrotide prophylaxis arm vs standard of care arm for the prevention of aGvHD.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥1 year of age at screening and undergoing allogeneic Hematopoietic Stem Cell Transplant (HSCT).
2. Participant must be diagnosed with acute leukemia in morphologic complete remission (CR1 or CR2) or with Myelodysplastic syndrome (MDS) with no circulating blasts and with less than 5% blasts in the bone marrow
3. Participant must have planned to receive either a myeloablative or reduced-intensity conditioning regimen and have an unrelated donor who is human leukocyte antigen (HLA) matched or single-allele mismatched
4. Participant must receive the following medical regimen as part of standard of care immunoprophylaxis for GvHD in either study arm at doses and regimen determined by local institutional guidelines, physician preference, and participant need:

   Methotrexate (MTX) or Mycophenolate mofetil (MMF) + calcineurin inhibitor (Cyclosporine A [CSA] or Tacrolimus [TAC]) +/- Anti-thymocyte globulin (ATG) (ATG use is limited to 30% of participants).
5. Graft must be a CD3+ T-cell replete peripheral blood stem cell (PBSC) graft or non-manipulated bone marrow (BM) graft.
6. Adult participants must be able to understand and sign a written informed consent. For pediatric participants, the parent/legal guardian or representative must be able to understand and sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines.

Exclusion Criteria:

1. Participant has had a prior autologous or allogeneic HSCT.
2. Participant is using or plans to use an investigational agent for the prevention of GvHD.
3. Participant is receiving or plans to receive other investigational therapy and/or is enrolled or plans to enroll in a separate clinical study.
4. Participant, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
5. Participant has a psychiatric illness that would prevent the participant or legal guardian or representative from giving informed consent and/or assent.
6. Participant has a serious active disease or co-morbid medical condition, as judged by the investigator, which would interfere with the conduct of this study.
7. Participant is pregnant or lactating and does not agree to stop breastfeeding.
8. Any other condition that would cause a risk to the participant if he/she participated in the trial.
9. Participant has a known history of hypersensitivity to defibrotide or any of the excipients.
10. Participant had acute bleeding that is clinically significant within 24 hours before the start of study treatment, defined as either of the following:

    * Hemorrhage requiring >15 cc/kg of packed red blood cells (eg, pediatric participant weighing 20 kg and requiring 300 cc packed red blood cells/24 hours, or an adult weighing >70 kg and requiring 3 units of packed red blood cells/24hours) to replace blood loss, or
    * Bleeding from a site which, in the investigator's opinion, constituted a potential life-threatening source (eg, pulmonary hemorrhage or central nervous system bleeding), irrespective of amount of blood loss
11. Participant used any medication that increases the risk of bleeding within 24 hours before the start of study treatment, including, but not limited to, systemic heparin, low molecular weight heparin, heparin analogs, alteplase, streptokinase, urokinase, antithrombin III, oral anticoagulants including warfarin, and other agents that increase the risk of bleeding. Participants may have received heparin or other anticoagulants for routine central venous line management and intermittent dialysis or ultrafiltration. Fibrinolytic instillation for central venous line occlusion was also permitted. Note: Heparin used to keep catheters open was allowed (up to 100 U/kg/day).

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (62):
- United States (18):
  - USC Norris Cancer Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - Mayo Clinic Jacksonville - PPDS, Jacksonville, Florida
  - Blood & Marrow Transplant Center, Orlando, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Kansas Medical Center, Westwood, Kansas
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Montefiore Einstein Cancer Center, The Bronx, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - MUSC-Hollings Cancer Center, Charleston, South Carolina
  - VA Puget Sound Health Care System, Seattle, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
- Austria (2):
  - Universitätsklinikum Innsbruck, Innsbruck
  - Ordensklinikum Linz, Krankenhaus der Elisabethinen GmbH, Linz
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Gent, Ghent
  - UZ Leuven, Leuven
- Specialized Hospital for Active Treatment of Haematological Diseases - Sofia, Sofia, Bulgaria
- Canada (3):
  - Hôpital Maisonneuve-Rosemont, Montreal
  - Sainte Justine Hospital, Montreal
  - McGill University Health Center, Montreal
- Klinichki Bolnicki Centar Zagreb, Zagreb, Croatia
- France (4):
  - Hospital d Instructions des Armees Percy, Clamart
  - CHRU Lille, Lille
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (11):
  - Helios Klinikum Berlin Buch, Berlin
  - Medizinische Universitätsklinik Knappschaftskrankenhaus, Bochum
  - Klinikum Frankfurt (Oder) GmbH, Brandenburg
  - Uniklinik Köln, Cologne
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - University Medicine Göttingen Germany, Göttingen
  - Universitaetsklinikum Halle (Saale), Halle
  - Universitatsklinikum Leipzig, Leipzig
  - Klinikum Mannheim Universitätsklinikum gGmbH, Mannheim
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Klinikum der Universitat Regensburg, Regensburg
- Greece (2):
  - Attikon University General Hospital, Athens
  - University General Hospital of Patras, Pátrai
- Italy (3):
  - ASST Grande Ospedale Metropolitano Niguarda - Presidio Ospedaliero Ospedale Niguarda Ca' Granda, Milan
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Ospedale Pediatrico Bambino Gesù, Roma
- Poland (2):
  - Centrum Onkologii im. Marii Sklodowskiej-Curie, Warsaw
  - Dolnoslaskie Centrum Transplantacji Komorkowych z Krajowym Bankiem Dawcow Szpiku, Wroclaw
- Instituto Português de Oncologia de Lisboa Francisco Gentil, E.P.E., Lisbon, Portugal
- Spain (6):
  - Hospital Universitario Marques de Valdecilla, A Coruña
  - Hospital de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
  - Complejo Asistencial Universitario de Salamanca - H. Clinico, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (5):
  - Birmingham Heartlands Hospital, Birmingham
  - St James University Hospital, Leeds
  - St. James University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Manchester Royal Infirmary, Manchester

REFERENCES:
- [Derived] Hudspeth M, Mori S, Nachbaur D, Perez-Simon JA, Stolzel F, Riches M, Wu W, Zhang P, Agarwal S, Yakoub-Agha I. A phase II, prospective, randomized, open-label study of defibrotide added to standard-of-care prophylaxis for the prevention of acute graft-versus-host disease after allogeneic hematopoietic cell transplantation. Haematologica. 2023 Apr 1;108(4):1026-1038. doi: 10.3324/haematol.2022.281471. PMID 36519326

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Informed Consent and/or assent was obtained from participants, parents/legal guardians or representatives.
Groups:
- Defibrotide Prophylaxis: Participants were administered Defibrotide Prophylaxis solution intravenously by study personnel at a dose of 25 mg/kg/day (6.25 mg/kg via 2-hour IV infusion every 6 hours) and Standard of Care immunoprophylaxis according to local institutional guidelines, physician preference, and patient need.
- Standard of Care Immunoprophylaxis: Participants were administered Standard of Care immunoprophylaxis alone according to local institutional guidelines, physician preference, and patient need.
Period: Overall Study
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Started | 79 | 73
Completed | 56 | 59
Not Completed | 23 | 14
Not completed — Relapse of Hematologic Disease | 1 | 0
Not completed — Death | 10 | 7
Not completed — Hepatic Candidosis | 1 | 0
Not completed — Adverse Event, Serious Fatal | 0 | 2
Not completed — Consent Withdrawn by Participant | 3 | 3
Not completed — Disease Relapse | 2 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Relapse of Disease New Transplant Performed | 1 | 0
Not completed — Problems with Donor and Diagnosis of Early Relapse | 1 | 0
Not completed — Early Termination, Did Not Proceed to Transplant | 1 | 0
Not completed — Adverse Event, Non-fatal | 1 | 0
Not completed — Patient Relapsed and Did Not Proceed to Transplant | 0 | 1
Not completed — Patient Was Not Eligible | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed using the Intent-to-Treat (ITT) Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis | Total
Number analyzed (Participants) | 79 | 73 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.54 (16.952) | 51.09 (16.621) | 50.80 (16.741)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 37 | 75
  Male | 41 | 36 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 67 | 63 | 130
  Unknown or Not Reported | 11 | 9 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 66 | 63 | 129
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence Percentage of Grade B to D Acute Graft Versus Host Disease (aGvHD) by Day +100 Post-Hematopoietic Stem Cell Transplant (HSCT)
Description: Cumulative Incidence Percentage of Grade B to D aGvHD was defined using the International Bone Marrow Transplant Registry (IBMTR) Severity Index. Grade B is defined as Skin stage = 2 or Liver stage = 1 to 2 or GI stage = 1 to 2. Grade C is defined as Skin stage = 3 or Liver stage = 3 or GI stage = 3. Grade D is defined as a Skin stage = 4 or Liver stage = 4 or GI stage = 4.
Time Frame: HSCT Day (Day +0 post-HSCT) through Day +100 post-HSCT
Population: Cumulative Incidence Rate of Grade B to D Acute Graft Versus Host Disease (aGvHD) was assessed using the Intent-to-Treat Analysis Set.
Measure: Number; unit: cumulative incidence percentage
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 79 | 73
cumulative incidence percentage | 38.4 | 47.1

2. Secondary Outcome: Cumulative Incidence Percentage of Grade B to D aGvHD by Day +180 Post-HSCT
Description: Cumulative Incidence Percentage of Grade B to D aGvHD was defined using the IBMTR Severity Index. Grade B is defined as Skin stage = 2 or Liver stage = 1 to 2 or GI stage = 1 to 2. Grade C is defined as Skin stage = 3 or Liver stage = 3 or GI stage = 3. Grade D is defined as a Skin stage = 4 or Liver stage = 4 or GI stage = 4.
Time Frame: HSCT Day (Day +0 post-HSCT) through Day +180 post-HSCT
Population: as for outcome 1
Measure: Number; unit: cumulative incidence percentage
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 79 | 73
cumulative incidence percentage | 50.6 | 51.6

3. Secondary Outcome: Kaplan-Meier Estimate of Grade B to D aGvHD-free Survival by Days +100 and +180 Post-HSCT
Description: Grade B to D aGvHD was defined using the IBMTR Severity Index. Grade B is defined as Skin stage = 2 or Liver stage = 1 to 2 or GI stage = 1 to 2. Grade C is defined as Skin stage = 3 or Liver stage = 3 or GI stage = 3. Grade D is defined as a Skin stage = 4 or Liver stage = 4 or GI stage = 4.
Time Frame: HSCT Day (Day +0 post-HSCT) through Days +100 and +180 post-HSCT
Population: Kaplan-Meier Estimate of Grade B to D aGvHD-free Survival was assessed using the Intent-to-Treat Analysis Set.
Measure: Number; unit: percentage of participants
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 79 | 73
percentage of participants
  Day +100 post-HSCT | 60.3 | 51.4
  Day +180 post-HSCT | 45.1 | 42.6

4. Secondary Outcome: Cumulative Incidence Percentage of Grade C to D aGvHD by Days +100 and +180 Post-HSCT
Description: Cumulative Incidence Percentage of Grade C to D aGvHD was defined using the IBMTR Severity Index. Grade C is defined as Skin stage = 3 or Liver stage = 3 or GI stage = 3. Grade D is defined as a Skin stage = 4 or Liver stage = 4 or GI stage = 4.
Time Frame: HSCT Day (Day +0 post-HSCT) through Days +100 and +180 post-HSCT
Population: Cumulative Incidence Rate of Grade C to D Acute Graft Versus Host Disease (aGvHD) was assessed using the Intent-to-Treat Analysis Set.
Measure: Number; unit: cumulative incidence percentage
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 79 | 73
cumulative incidence percentage
  Day +100 post-HSCT | 16.5 | 21.5
  Day +180 post-HSCT | 22.7 | 25.9

5. Secondary Outcome: Cumulative Incidence Percentage of Disease Relapse by Days +100 and +180 Post-HSCT
Description: Disease relapse was defined by either morphological evidence of acute leukemia or Myelodysplastic syndrome (MDS) consistent with pre-transplant features, documented or not by biopsy. The event was defined as an increase in size of prior sites of disease or evidence of new sites of disease, documented or not by biopsy. Disease relapse was diagnosed when there was morphological or clinical evidence of the following: reappearance of leukemia blast cells in the peripheral blood, or >5% blasts in the bone marrow (BM), not attributable to another cause (eg, BM regeneration), or the appearance of previous or new dysplastic changes (MDS specific) within the BM, with or without falling donor chimerism, or the development of extramedullary leukemia or leukemic cells in the cerebral spinal fluid, or institution of therapy to treat relapsed disease, including donor lymphocyte infusion.
Time Frame: HSCT Day (Day +0 post-HSCT) through Days +100 and +180 post-HSCT
Population: Cumulative Incidence Rate of Disease Relapse was assessed using the Intent-to-Treat Analysis Set.
Measure: Number; unit: cumulative incidence percentage
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 79 | 73
cumulative incidence percentage
  Day +100 post-HSCT | 11.0 | 4.3
  Day +180 post-HSCT | 16.8 | 5.8

6. Secondary Outcome: Cumulative Incidence Percentage of Systemic Steroids for the Treatment of aGvHD +180 Days Post-HSCT
Description: For each treatment arm, the cumulative incidence rate of systemic steroid use for the treatment of aGvHD by Day +180 post-HSCT will be estimated using the cumulative incidence competing risk estimator. The calculation of the cumulative incidence rates and the stratified Gray's test was carried out using the LIFETEST procedure in SAS version 9.4. If the participant experienced a competing risk event, then the initiation date was used to calculate the time-to-event variable.
Time Frame: HSCT Day (Day +0 post-HSCT) through Day +180 post-HSCT
Population: Cumulative Incidence Rate of Systemic Steroids for the Treatment of aGvHD was assessed using the Intent-to-Treat Analysis Set.
Measure: Number; unit: cumulative incidence percentage
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 79 | 73
cumulative incidence percentage | 38.2 | 28.6

7. Secondary Outcome: Change From Baseline to Days +100 and +180 Post-HSCT in the Physical Wellbeing Subscale as Measured by the Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) Questionnaire Score
Description: The Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) total score is the sum of the FACT physical wellbeing score, the FACT social/family wellbeing score, the FACT emotional wellbeing score, the FACT functional wellbeing score, and the FACT-BMT subscale. The FACT physical wellbeing subscale scores range from a minimum of 0 to a maximum of 28, with higher scores indicating better quality of life. A negative change from baseline indicates a decrease in score.
Time Frame: Baseline through Days +100 and +180 post-HSCT
Population: Only participants with age >=16 years at baseline in the Safety Analysis Set were used in this analysis.
Measure: Mean (Standard Deviation); unit: unit on a scale
Groups:
- Standard of Care Immunoprohylaxis: Participants were administered Standard of Care immunoprophylaxis alone according to local institutional guidelines, physician preference, and patient need.
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprohylaxis
Number analyzed (Participants) | 70 | 67
unit on a scale
  Change from Baseline to Day +100 post-HSCT | -1.25 (5.069) | -1.41 (6.371)
  Change from Baseline to Day +180 post-HSCT | -1.55 (5.230) | -1.54 (5.717)

8. Secondary Outcome: Change From Baseline to Days +100 and +180 Post-HSCT in the Social/Family Wellbeing Subscale as Measured by the FACT-BMT Questionnaire Score
Description: The Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) total score is the sum of the FACT physical wellbeing score, the FACT social/family wellbeing score, the FACT emotional wellbeing score, the FACT functional wellbeing score, and the FACT-BMT subscale. The FACT social/family wellbeing subscale scores range from a minimum of 0 to a maximum of 28, with higher scores indicating better quality of life. A negative change from baseline indicates a decrease in score.
Time Frame: Baseline through Days +100 and +180 post-HSCT
Population: Only participants with age >=16 years at baseline in the Safety Analysis Set were used in this analysis.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 70 | 67
unit on a scale
  Change from Baseline to Day +100 post-HSCT | -0.56 (3.488) | -0.29 (5.716)
  Change from Baseline to Day +180 post-HSCT | -0.78 (4.085) | -1.34 (3.380)

9. Secondary Outcome: Change From Baseline to Days +100 and +180 Post-HSCT in the Emotional Wellbeing Subscale as Measured by the FACT-BMT Questionnaire Score
Description: The Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) total score is the sum of the FACT physical wellbeing score, the FACT social/family wellbeing score, the FACT emotional wellbeing score, the FACT functional wellbeing score, and the FACT-BMT subscale. The FACT emotional wellbeing subscale scores range from a minimum of 0 to a maximum of 24, with higher scores indicating better quality of life.
Time Frame: Baseline through Days +100 and +180 post-HSCT
Population: Only participants with age >=16 years at baseline in the Safety Analysis Set were used in this analysis.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 70 | 67
unit on a scale
  Change from Baseline to Day +100 post-HSCT | 1.47 (4.910) | 1.47 (3.659)
  Change from Baseline to Day +180 post-HSCT | 0.79 (4.683) | 1.53 (3.458)

10. Secondary Outcome: Change From Baseline to Days +100 and +180 Post-HSCT in the Functional Wellbeing Subscale as Measured by the FACT-BMT Questionnaire Score
Description: The Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) total score is the sum of the FACT physical wellbeing score, the FACT social/family wellbeing score, the FACT emotional wellbeing score, the FACT functional wellbeing score, and the FACT-BMT subscale. The FACT functional wellbeing subscale scores range from a minimum of 0 to a maximum of 28, with higher scores indicating better quality of life. A negative change from baseline indicates a decrease in score.
Time Frame: Baseline through Days +100 and +180 post HSCT
Population: Only participants with age >=16 years at baseline in the Safety Analysis Set were used in this analysis.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 70 | 67
unit on a scale
  Change from Baseline to Day +100 post-HSCT | -1.71 (5.622) | -2.11 (5.962)
  Change from Baseline to Day +180 post-HSCT | -2.21 (7.241) | -0.95 (6.627)

11. Secondary Outcome: Change From Baseline to Days +100 and +180 Post-HSCT in the Bone Marrow Transplantation Subscale (BMTS) as Measured by the FACT-BMT Questionnaire Score
Description: The Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) total score is the sum of the FACT physical wellbeing score, the FACT social/family wellbeing score, the FACT emotional wellbeing score, the FACT functional wellbeing score, and the FACT-BMT subscale. The FACT-BMT subscale scores range from a minimum of 0 to a maximum of 40, with higher scores indicating better quality of life. A negative change from baseline indicates a decrease in score.
Time Frame: Baseline through Days +100 and +180 post-HSCT
Population: Only participants with age >=16 years at baseline in the Safety Analysis Set were used in this analysis.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 70 | 67
unit on a scale
  Change from Baseline to Day +100 post-HSCT | -0.88 (5.484) | -2.14 (5.900)
  Change from Baseline to Day +180 post-HSCT | -2.33 (7.037) | -1.01 (6.173)

12. Secondary Outcome: Change From Baseline to Days +100 and +180 Post-HSCT in the General (FACT-G) Questionnaire Score
Description: The FACT-General (FACT-G) is a core component of the FACT-BMT, and includes 4 of the 5 subscales included in the FACT-BMT total score (FACT physical wellbeing score, FACT social/family wellbeing score, FACT emotional wellbeing score, the FACT functional wellbeing score). In line with this similarity, results of the FACT-G exhibited the same pattern as described for the FACT-BMT total score. The FACT-G scores range from a minimParticipants were age ≥16 years at baseline.
Time Frame: Baseline through Days +100 and +180 post-HSCT
Population: Only participants with age >=16 years at baseline in the Safety Analysis Set were used in this analysis.
Measure: Mean (Standard Deviation); unit: unit on a scale
Groups:
- Standard of Care Immunoprophylaxis: Participants were administered Standard of Care immunoprophylaxis alone in a 1:1 ratio according to local institutional guidelines, physician preference, and patient need.
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 70 | 67
unit on a scale
  Change from Baseline to Day +100 post-HSCT | -2.38 (12.623) | -1.74 (15.623)
  Change from Baseline to Day +180 post-HSCT | -4.03 (15.366) | -1.33 (13.613)

13. Secondary Outcome: Change From Baseline to Days +100 and +180 Post-HSCT in the FACT-BMT Total Score
Description: The Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) total score is the sum of the FACT physical wellbeing score, the FACT social/family wellbeing score, the FACT emotional wellbeing score, the FACT functional wellbeing score, and the FACT-BMT subscale. The FACT-BMT total score range is from a minimum of 0 to a maximum of 148, with higher scores indicating better quality of life. A negative change from baseline indicates a decrease in score.
Time Frame: Baseline through Days +100 and +180 post-HSCT
Population: Only participants with age >=16 years at baseline in the Safety Analysis Set were used in this analysis.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 70 | 67
unit on a scale
  Change from Baseline to Day +100 post-HSCT | -3.24 (16.036) | -3.70 (19.854)
  Change from Baseline to Day +180 post-HSCT | -6.38 (21.358) | -2.83 (18.079)

14. Secondary Outcome: Change From Baseline to Days +100 and +180 Post-HSCT in the Functional Assessment of Cancer Therapy-Bone Marrow Transplant-Trial Outcomes Index (FACT-BMT-TOI)
Description: The FACT-BMT-TOI is defined as the sum of the FACT physical wellbeing score, the FACT functional wellbeing score, and the FACT-BMT subscale. Scores range from a minimum of 0 to a maximum of 96, with higher scores indicating better quality of life. A negative change from baseline indicates a decrease in score.
Time Frame: Baseline through Days +100 and +180 post-HSCT
Population: Only participants with age >=16 years at baseline in the Safety Analysis Set were used in this analysis.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 70 | 67
unit on a scale
  Change from Baseline to Day +100 post-HSCT | -3.88 (13.110) | -5.24 (15.575)
  Change from Baseline to Day +180 post-HSCT | -6.99 (17.393) | -3.33 (14.922)

15. Secondary Outcome: Change From Baseline to Days +100 and +180 Post-HSCT in Participant Reported Outcomes Measured Based on the EQ-5D-5L Index Value for Health States
Description: The 5-Level EuroQol-5D health questionnaire (EQ-5D-5L) index value, which is country-specific, was only performed for participants in the US. The EQ-5D-5L is a standardized instrument for use as a measure of health outcome that includes a descriptive system consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Change from the baseline assessment to Days +100 and +180 post-HSCT in the index value was assessed. The index value total range is from a minimum value of -1 to a maximum value of +1. A higher EQ-5D-5L index value represents better quality of life (QoL), thus a positive change in the index value represents improved QoL.
Time Frame: Baseline through Days +100 and +180 post-HSCT
Population: Only participants with age >=16 years at baseline in the Safety Analysis Set were used in this analysis.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 70 | 67
unit on a scale
  Change from Baseline to Day +100 post-HSCT | 0.02 (0.092) | -0.01 (0.101)
  Change from Baseline to Day +180 post-HSCT | 0.02 (0.078) | -0.01 (0.121)

16. Secondary Outcome: Change From Baseline to Days +100 and +180 Post-HSCT in Participant Reported Outcomes as Measured Based on the EQ Visual Analog Scale (EQ VAS)
Description: The EQ VAS score at baseline and each of the post-HSCT assessments was summarized and presented using descriptive statistics. A higher EQ VAS score represents better QoL. For each of the post-HSCT assessments, change between baseline and that assessment in the EQ VAS score was calculated similarly to the EQ-5D-5L index value for a specific participant and was summarized and presented using descriptive statistics. The score ranges from a minimum of 0 and a maximum of 100. A negative change in the score indicates a decrease in quality of life.
Time Frame: Baseline through Days +100 and +180 post-HSCT
Population: Only participants with age >=16 years at baseline in the Safety Analysis Set were used in this analysis.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 70 | 67
unit on a scale
  Change from Baseline to Day +100 post-HSCT | 6.03 (20.599) | 2.70 (15.004)
  Change from Baseline to Day +180 post-HSCT | 2.24 (29.023) | -0.90 (21.530)

17. Secondary Outcome: Change From Baseline to Day +100 Post-HSCT in 5-Level European Quality of Life (EQ-5D-5L) Mobility Dimension for Participants With Age >=16 Years
Description: The EQ-5D-5L is a standardized instrument for use as a measure of health outcome that includes a descriptive system consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each of the 5 dimensions based on the descriptive system of the EQ-5D-5L, the numbers of participants for all categories (the 5 levels of reported problems) were assessed. For Day +100 Post-HSCT change between baseline in each dimension will be categorized as follows for a specific participant: Condition improved, if the reported level of problem is lower at that assessment than at baseline; Condition unchanged, if the reported level of problem remains the same; Condition deteriorated, if the reported level of problem is higher at that assessment than at baseline; Unknown, if the reported level of problem is not completed or missing either at baseline or at that assessment.
Time Frame: Baseline through Day +100 post-HSCT
Population: Only participants with age >=16 years at baseline in the Safety Analysis Set who were on the study at the time of the scheduled post-baseline assessment were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 61 | 62
Participants
  Condition improved | 3 | 4
  Condition unchanged | 31 | 28
  Condition deteriorated | 8 | 15
  Unknown | 19 | 15

18. Secondary Outcome: Change From Baseline to Day +180 Post-HSCT in 5-Level European Quality of Life (EQ-5D-5L) Mobility Dimension for Participants With Age >=16 Years
Description: The EQ-5D-5L is a standardized instrument for use as a measure of health outcome that includes a descriptive system consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each of the 5 dimensions based on the descriptive system of the EQ-5D-5L, the numbers of participants for all categories (the 5 levels of reported problems) were assessed. For Day +180 Post-HSCT change between baseline in each dimension will be categorized as follows for a specific participant: Condition improved, if the reported level of problem is lower at that assessment than at baseline; Condition unchanged, if the reported level of problem remains the same; Condition deteriorated, if the reported level of problem is higher at that assessment than at baseline; Unknown, if the reported level of problem is not completed or missing either at baseline or at that assessment.
Time Frame: Baseline through Day +180 post-HSCT
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 57 | 61
Participants
  Condition improved | 3 | 3
  Condition unchanged | 26 | 25
  Condition deteriorated | 11 | 14
  Unknown | 17 | 19

19. Secondary Outcome: Change From Baseline to Day +100 Post-HSCT in 5-Level European Quality of Life (EQ-5D-5L) Pain/Discomfort Dimension for Participants With Age >=16 Years
Description: The EQ-5D-5L is a standardized instrument for use as a measure of health outcome that includes a descriptive system consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each of the 5 dimensions based on the descriptive system of the EQ-5D-5L, the numbers of participants for all categories (the 5 levels of reported problems) were assessed. For Days +100 Post-HSCT change between baseline in each dimension will be categorized as follows for a specific participant: Condition improved, if the reported level of problem is lower at that assessment than at baseline; Condition unchanged, if the reported level of problem remains the same; Condition deteriorated, if the reported level of problem is higher at that assessment than at baseline; Unknown, if the reported level of problem is not completed or missing either at baseline or at that assessment.
Time Frame: Baseline through Day +100 post-HSCT
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 61 | 62
Participants
  Condition improved | 10 | 9
  Condition unchanged | 18 | 20
  Condition deteriorated | 14 | 18
  Unknown | 19 | 15

20. Secondary Outcome: Change From Baseline to Day +180 Post-HSCT in 5-Level European Quality of Life (EQ-5D-5L) Pain/Discomfort Dimension for Participants With Age >=16 Years
Description: as for outcome 18
Time Frame: Baseline through Day +180 post-HSCT
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 57 | 61
Participants
  Condition improved | 6 | 8
  Condition unchanged | 23 | 20
  Condition deteriorated | 11 | 14
  Unknown | 17 | 19

21. Secondary Outcome: Change From Baseline to Day +100 Post-HSCT in 5-Level European Quality of Life (EQ-5D-5L) Self-Care Dimension for Participants With Age >=16 Years
Description: as for outcome 17
Time Frame: Baseline through Day +100 post-HSCT
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 61 | 62
Participants
  Condition improved | 1 | 0
  Condition unchanged | 34 | 37
  Condition deteriorated | 7 | 10
  Unknown | 19 | 15

22. Secondary Outcome: Change From Baseline to Day +180 Post-HSCT in 5-Level European Quality of Life (EQ-5D-5L) Self-Care Dimension for Participants With Age >=16 Years
Description: as for outcome 18
Time Frame: Baseline through Day +180 post-HSCT
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 57 | 61
Participants
  Condition improved | 2 | 1
  Condition unchanged | 34 | 31
  Condition deteriorated | 4 | 10
  Unknown | 17 | 19

23. Secondary Outcome: Change From Baseline to Day +100 Post-HSCT in 5-Level European Quality of Life (EQ-5D-5L) Usual Activities Dimension for Participants With Age >=16 Years
Description: as for outcome 17
Time Frame: Baseline through Day +100 post-HSCT
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 61 | 62
Participants
  Condition improved | 8 | 7
  Condition unchanged | 21 | 22
  Condition deteriorated | 13 | 18
  Unknown | 19 | 15

24. Secondary Outcome: Change From Baseline to Day +180 Post-HSCT in 5-Level European Quality of Life (EQ-5D-5L) Usual Activities Dimension for Participants With Age >=16 Years
Description: as for outcome 18
Time Frame: Baseline through Day +180 post-HSCT
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 57 | 61
Participants
  Condition improved | 10 | 5
  Condition unchanged | 16 | 19
  Condition deteriorated | 14 | 18
  Unknown | 17 | 19

25. Secondary Outcome: Change From Baseline to Day +100 Post-HSCT in 5-Level European Quality of Life (EQ-5D-5L) Anxiety/Depression Dimension for Participants With Age >=16 Years
Description: as for outcome 17
Time Frame: Baseline through Day +100 post-HSCT
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 61 | 62
Participants
  Condition improved | 7 | 10
  Condition unchanged | 27 | 30
  Condition deteriorated | 8 | 7
  Unknown | 19 | 15

26. Secondary Outcome: Change From Baseline to Day +180 Post-HSCT in 5-Level European Quality of Life (EQ-5D-5L) Anxiety/Depression Dimension for Participants With Age >=16 Years
Description: as for outcome 18
Time Frame: Baseline through Day +180 post-HSCT
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
Number analyzed (Participants) | 57 | 61
Participants
  Condition improved | 8 | 12
  Condition unchanged | 21 | 23
  Condition deteriorated | 11 | 6
  Unknown | 17 | 20

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) and Serious Adverse Events (SAEs) were reported from the time of signed informed consent form (ICF) and were recorded up to Day +63 post-HSCT. SAEs considered by the investigator to be related to study drug or study procedures were reported up to Day +180 post-HSCT.
Description: Treatment-emergent adverse events (TEAEs) were defined as events that occurred after randomization into this study. A TEAE is defined as any event with a start date on or after baseline through the end of the study, or any ongoing event that worsens in severity after baseline through the end of the study. Adverse events were assessed using the Safety Analysis Set.
Arm/Group | Defibrotide Prophylaxis | Standard of Care Immunoprophylaxis
All-Cause Mortality (participants affected / at risk) | 10/74 | 9/70
Serious Adverse Events (participants affected / at risk) | 31/74 | 31/70
Other Adverse Events (participants affected / at risk) | 74/74 | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Defibrotide Prophylaxis (N=74) | Standard of Care Immunoprophylaxis (N=70)
Obstructive shock (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 1
Venoocclusive disease (Vascular disorders) | 1 | 1
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Epstein-Barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute graft versus host disease (Immune system disorders) | 4 | 1
Acute graft versus host disease in skin (Immune system disorders) | 1 | 4
Graft versus host disease (Immune system disorders) | 0 | 1
Graft versus host disease in liver (Immune system disorders) | 0 | 1
Acute graft versus host disease in intestine (Immune system disorders) | 2 | 1
General physical health deterioration (General disorders) | 0 | 1
Mucosal haemorrhage (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (General disorders) | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Evans syndrome (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Venoocclusive liver disease (Hepatobiliary disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 3 | 2
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 1
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cystitis viral (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Cytomegalovirus viraemia (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Epstein-Barr viraemia (Infections and infestations) | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0
Fungaemia (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Septic shock (Infections and infestations) | 0 | 2
Serratia infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Defibrotide Prophylaxis (N=74) | Standard of Care Immunoprophylaxis (N=70)
Flushing (Vascular disorders) | 4 | 4
Hypertension (Vascular disorders) | 25 | 29
Hypotension (Vascular disorders) | 13 | 11
Orthostatic hypotension (Vascular disorders) | 6 | 3
Graft versus host disease in skin (Immune system disorders) | 4 | 2
Asthenia (General disorders) | 9 | 6
Catheter site pain (General disorders) | 8 | 9
Chills (General disorders) | 7 | 6
Fatigue (General disorders) | 25 | 25
Mucosal inflammation (General disorders) | 10 | 17
Oedema peripheral (General disorders) | 19 | 21
Pain (General disorders) | 5 | 6
Pyrexia (General disorders) | 28 | 24
Agitation (Psychiatric disorders) | 5 | 3
Anxiety (Psychiatric disorders) | 11 | 9
Confusional state (Psychiatric disorders) | 5 | 3
Delirium (Psychiatric disorders) | 4 | 2
Depression (Psychiatric disorders) | 7 | 2
Insomnia (Psychiatric disorders) | 22 | 16
Fall (Injury, poisoning and procedural complications) | 5 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 6
Limb injury (Injury, poisoning and procedural complications) | 4 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 4
Alanine aminotransferase increased (Investigations) | 3 | 7
Aspartate aminotransferase increased (Investigations) | 2 | 5
Bacterial test positive (Investigations) | 4 | 3
Blood bilirubin increased (Investigations) | 3 | 5
Blood creatinine increased (Investigations) | 12 | 6
Blood magnesium decreased (Investigations) | 1 | 4
C-reactive protein increased (Investigations) | 4 | 5
Epstein-Barr virus test positive (Investigations) | 4 | 2
Neutrophil count decreased (Investigations) | 8 | 11
Platelet count decreased (Investigations) | 19 | 21
Transaminases increased (Investigations) | 4 | 6
Weight decreased (Investigations) | 3 | 4
White blood cell count decreased (Investigations) | 8 | 6
Sinus tachycardia (Cardiac disorders) | 9 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 11
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 12
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Anaemia (Blood and lymphatic system disorders) | 27 | 30
Febrile neutropenia (Blood and lymphatic system disorders) | 30 | 20
Leukopenia (Blood and lymphatic system disorders) | 9 | 6
Neutropenia (Blood and lymphatic system disorders) | 12 | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 19 | 19
Dizziness (Nervous system disorders) | 10 | 8
Dysgeusia (Nervous system disorders) | 10 | 9
Headache (Nervous system disorders) | 31 | 23
Restless legs syndrome (Nervous system disorders) | 5 | 1
Somnolence (Nervous system disorders) | 5 | 2
Tremor (Nervous system disorders) | 10 | 9
Dry eye (Eye disorders) | 15 | 6
Eye swelling (Eye disorders) | 0 | 4
Abdominal distension (Gastrointestinal disorders) | 8 | 5
Abdominal pain (Gastrointestinal disorders) | 13 | 22
Abdominal pain lower (Gastrointestinal disorders) | 4 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 9
Constipation (Gastrointestinal disorders) | 28 | 29
Diarrhoea (Gastrointestinal disorders) | 47 | 53
Dry mouth (Gastrointestinal disorders) | 7 | 6
Dyspepsia (Gastrointestinal disorders) | 4 | 11
Dysphagia (Gastrointestinal disorders) | 5 | 3
Flatulence (Gastrointestinal disorders) | 4 | 3
Haemorrhoids (Gastrointestinal disorders) | 6 | 6
Mouth ulceration (Gastrointestinal disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 56 | 49
Odynophagia (Gastrointestinal disorders) | 7 | 3
Oesophagitis (Gastrointestinal disorders) | 5 | 0
Stomatitis (Gastrointestinal disorders) | 42 | 36
Vomiting (Gastrointestinal disorders) | 39 | 38
Acute kidney injury (Renal and urinary disorders) | 17 | 16
Cystitis haemorrhagic (Renal and urinary disorders) | 2 | 4
Dysuria (Renal and urinary disorders) | 6 | 5
Haematuria (Renal and urinary disorders) | 3 | 4
Pollakiuria (Renal and urinary disorders) | 4 | 4
Urinary retention (Renal and urinary disorders) | 4 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 8
Erythema (Skin and subcutaneous tissue disorders) | 13 | 13
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 2 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 13
Pruritus generalised (Skin and subcutaneous tissue disorders) | 4 | 5
Rash (Skin and subcutaneous tissue disorders) | 17 | 19
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 7
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 3
Decreased appetite (Metabolism and nutrition disorders) | 30 | 30
Dehydration (Metabolism and nutrition disorders) | 4 | 5
Fluid overload (Metabolism and nutrition disorders) | 5 | 5
Fluid retention (Metabolism and nutrition disorders) | 6 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 8
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 24 | 27
Hypomagnesaemia (Metabolism and nutrition disorders) | 30 | 35
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 5
Hypophagia (Metabolism and nutrition disorders) | 1 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 11
Malnutrition (Metabolism and nutrition disorders) | 4 | 6
Clostridium difficile colitis (Infections and infestations) | 3 | 4
Cytomegalovirus infection (Infections and infestations) | 11 | 14
Oral candidiasis (Infections and infestations) | 0 | 6
Urinary tract infection (Infections and infestations) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review trial results communications prior to public release and can embargo such communications for a period of at least 60 days from the time submitted to sponsor for review. If requested by sponsor, the PI will withhold publication for up to an additional 30 days. Furthermore, the first publication of study results must be a joint publication of all study sites unless a joint manuscript has not been submitted for publication within 12 months of completion of the study.

DOCUMENTS (2):
  • Study Protocol (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT03339297/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT03339297/SAP_001.pdf